CLINICAL TRIAL: NCT02083302
Title: Experimentally Testing the Effectiveness of a Campus-based Bystander Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-412M; 1R01CE001855-01 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-11 (Estimated); Last update posted 2014-03-11 (Estimated); Status verified 2014-03

CONDITIONS: Assaultive Behavior; Violence; Sexual Assault and Rape; Helping Behavior
Keywords: campus sexual assault; bystander intervention
MeSH Terms: conditions — Helping Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment1 (Experimental): The Treatment1 group received SCREAM Theater Dose 1, SCREAM Theater Dose 2 and SCREAM Theater Dose 3.
  Interventions: Behavioral: SCREAM Theater Dose 1; Behavioral: SCREAM Theater Doses 2 & SCREAM Theater Dose 3
- Treatment2 (Experimental): The Treatment2 group received SCREAM Theater Dose 1, SCREAM Theater Dose 2, SCREAM Theater Dose 3 and SCREAM Theater Dose 4.
  Interventions: Behavioral: SCREAM Theater Dose 1; Behavioral: SCREAM Theater Doses 2 & SCREAM Theater Dose 3; Behavioral: SCREAM Theater Dose 4
- Control (Other): The control group received SCREAM Theater Dose 1.
  Interventions: Behavioral: SCREAM Theater Dose 1

INTERVENTIONS:
Behavioral: SCREAM Theater Dose 1 — Intervention 1: A three part program: a skit acted out by peer educators that depicts a sexual assault; an in-character question and answer session; and an out-of-character information session.
Behavioral: SCREAM Theater Doses 2 & SCREAM Theater Dose 3 — Dose 2: Scenes from the skit from Session 1 are re-created with small groups of students, but stop at certain points to allow audience members to explore different bystander intervention possibilities.
  Dose 3: The six scenes outlined in Session 2 are presented individually to small groups of student participants; specifically outlining potential points of bystander intervention.
  Arms: Treatment1; Treatment2
Behavioral: SCREAM Theater Dose 4 — Booster Session
  Arms: Treatment2

SUMMARY:
The purpose of this study was to examine the impact of a bystander intervention education program on college students' attitudes and behaviors associated with bystander intervention and sexual violence.

DETAILED DESCRIPTION:
This study used a randomized control trial, longitudinal design to determine the impact of a peer education theater intervention on undergraduate student attitudes and behaviors related to sexual violence and bystander intervention. Students were assigned to either an experimental group (receiving 3-4 doses of the intervention ) or a comparison group (receiving 1 dose only) and were surveyed six times over an 18 month period.

ELIGIBILITY:
Inclusion Criteria:

* Incoming first year students in the fall semester of 2010
* Age 18 - 21
* Attended Summer Orientation session

Exclusion Criteria:

* Incoming transfer students
* Younger than 18 or older than 21

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4385 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Bystander Intentions | Change from baseline in bystander intentions to up to three months
  To measure intentions to be a bystander, we used the Bystander Attitude Scale, Revised (BAS-R) which is a modified version of Banyard's Bystander scale (Banyard, Plante, & Moynihan, 2005; see McMahon et al., in press, for scale development information). Participants were asked to indicate how likely they were to engage in the behavior in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Bystander Intentions | Change from baseline in bystander intentions to up to six months
  To measure intentions to be a bystander, we used the Bystander Attitude Scale, Revised (BAS-R) which is a modified version of Banyard's Bystander scale (Banyard, Plante, & Moynihan, 2005; see McMahon et al., in press, for scale development information). Participants were asked to indicate how likely they were to engage in the behavior in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Bystander Intentions | Change from baseline in bystander intentions to up to eight months
  To measure intentions to be a bystander, we used the Bystander Attitude Scale, Revised (BAS-R) which is a modified version of Banyard's Bystander scale (Banyard, Plante, & Moynihan, 2005; see McMahon et al., in press, for scale development information). Participants were asked to indicate how likely they were to engage in the behavior in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Bystander Intentions | Change from baseline in bystander intentions to up to fifteen months
  To measure intentions to be a bystander, we used the Bystander Attitude Scale, Revised (BAS-R) which is a modified version of Banyard's Bystander scale (Banyard, Plante, & Moynihan, 2005; see McMahon et al., in press, for scale development information). Participants were asked to indicate how likely they were to engage in the behavior in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Bystander Intentions | Change from baseline in bystander intentions to up to twenty months
  To measure intentions to be a bystander, we used the Bystander Attitude Scale, Revised (BAS-R) which is a modified version of Banyard's Bystander scale (Banyard, Plante, & Moynihan, 2005; see McMahon et al., in press, for scale development information). Participants were asked to indicate how likely they were to engage in the behavior in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.

SECONDARY OUTCOMES:
Bystander Friend Norms | Change from baseline in bystander friend norms to up to three months
  To measure friends' norms about being a bystander, we used the Bystander Attitude Scale, Revised (BAS-R). In this portion of the survey, participants were asked to indicate how likely they think their friends would be to engage in the items on the BAS-R in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely."Students' bystander friend norms were assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Bystander Friend Norms | Change from baseline in bystander friend norms to up to six months
  To measure friends' norms about being a bystander, we used the Bystander Attitude Scale, Revised (BAS-R). In this portion of the survey, participants were asked to indicate how likely they think their friends would be to engage in the items on the BAS-R in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander friend norms were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Bystander Friend Norms | Change from baseline in bystander friend norms to up to eight months
  To measure friends' norms about being a bystander, we used the Bystander Attitude Scale, Revised (BAS-R). In this portion of the survey, participants were asked to indicate how likely they think their friends would be to engage in the items on the BAS-R in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander friend norms were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Bystander Friend Norms | Change from baseline in bystander friend norms to up to fifteen months
  To measure friends' norms about being a bystander, we used the Bystander Attitude Scale, Revised (BAS-R). In this portion of the survey, participants were asked to indicate how likely they think their friends would be to engage in the items on the BAS-R in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander friend norms were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Bystander Friend Norms | Change from baseline in bystander friend norms to up to twenty months
  To measure friends' norms about being a bystander, we used the Bystander Attitude Scale, Revised (BAS-R). In this portion of the survey, participants were asked to indicate how likely they think their friends would be to engage in the items on the BAS-R in the future on a Likert scale from 1 - 5, "Unlikely" to "Very likely." Students' bystander friend norms were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.
Bystander Efficacy | Change from baseline in bystander efficacy to up to three months
  To assess level of confidence in one's ability to intervene, the Bystander Efficacy Scale was used (Banyard et al., 2007). Respondents were asked to rate their level of confidence that they would perform certain bystander behaviors on a scale of 0 ("can't do") to 100 ("very certain can do"). Students' bystander efficacy was assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Bystander Efficacy | Change from baseline in bystander efficacy to up to six months
  To assess level of confidence in one's ability to intervene, the Bystander Efficacy Scale was used (Banyard et al., 2007). Respondents were asked to rate their level of confidence that they would perform certain bystander behaviors on a scale of 0 ("can't do") to 100 ("very certain can do").Students' bystander efficacy was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Bystander Efficacy | Change from baseline in bystander efficacy to up to eight months
  To assess level of confidence in one's ability to intervene, the Bystander Efficacy Scale was used (Banyard et al., 2007). Respondents were asked to rate their level of confidence that they would perform certain bystander behaviors on a scale of 0 ("can't do") to 100 ("very certain can do"). Students' bystander efficacy was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Bystander Efficacy | Change from baseline in bystander efficacy to up to fifteen months
  To assess level of confidence in one's ability to intervene, the Bystander Efficacy Scale was used (Banyard et al., 2007). Respondents were asked to rate their level of confidence that they would perform certain bystander behaviors on a scale of 0 ("can't do") to 100 ("very certain can do"). Students' bystander efficacy was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Bystander Efficacy | Change from baseline in bystander efficacy to up to twenty months
  To assess level of confidence in one's ability to intervene, the Bystander Efficacy Scale was used (Banyard et al., 2007). Respondents were asked to rate their level of confidence that they would perform certain bystander behaviors on a scale of 0 ("can't do") to 100 ("very certain can do"). Students' bystander intentions were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.
Bystander Behavior | Change from baseline in bystander behavior to up to three months
  To measure actual bystander behavior, we used the Bystander Attitude Scale, Revised (BAS-R), which contains 18 items, each stating a different bystander behavior. For this portion of the survey, participants were asked whether they actually participated in the behavior in the previous month. Respondents can indicate "Yes", "No", or "Wasn't in the Situation".Students' bystander behavior was assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Bystander Behavior | Change from baseline in bystander behavior to up to six months
  To measure actual bystander behavior, we used the Bystander Attitude Scale, Revised (BAS-R), which contains 18 items, each stating a different bystander behavior. For this portion of the survey, participants were asked whether they actually participated in the behavior in the previous month. Respondents can indicate "Yes", "No", or "Wasn't in the Situation".Students' bystander behavior was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Bystander Behavior | Change from baseline in bystander behavior to up to eight months
  To measure actual bystander behavior, we used the Bystander Attitude Scale, Revised (BAS-R), which contains 18 items, each stating a different bystander behavior. For this portion of the survey, participants were asked whether they actually participated in the behavior in the previous month. Respondents can indicate "Yes", "No", or "Wasn't in the Situation". Students' bystander behavior was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Bystander Behavior | Change from baseline in bystander behavior to up to fifteen months
  To measure actual bystander behavior, we used the Bystander Attitude Scale, Revised (BAS-R), which contains 18 items, each stating a different bystander behavior. For this portion of the survey, participants were asked whether they actually participated in the behavior in the previous month. Respondents can indicate "Yes", "No", or "Wasn't in the Situation".Students' bystander behavior was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Bystander Behavior | Change from baseline in bystander behavior to up to twenty months
  To measure actual bystander behavior, we used the Bystander Attitude Scale, Revised (BAS-R), which contains 18 items, each stating a different bystander behavior. For this portion of the survey, participants were asked whether they actually participated in the behavior in the previous month. Respondents can indicate "Yes", "No", or "Wasn't in the Situation". Students' bystander behavior was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.
Rape Myth Acceptance | Change from baseline in rape myth acceptance to up to three months
  A revised version of the Illinois Rape Myth Acceptance Scale (Payne, Lonsway, & Fitzgerald, 1999) was used. The revised version (McMahon & Farmer, 2011) was selected because the scale includes updated language for college students as well as having a specific focus on accountability for rape and victim blaming (for information on scale development, see McMahon & Farmer, 2011). Students' rape myth acceptance was assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Rape Myth Acceptance | Change from baseline in rape myth acceptance to up to six months
  A revised version of the Illinois Rape Myth Acceptance Scale (Payne, Lonsway, & Fitzgerald, 1999) was used. The revised version (McMahon & Farmer, 2011) was selected because the scale includes updated language for college students as well as having a specific focus on accountability for rape and victim blaming (for information on scale development, see McMahon & Farmer, 2011).Students' rape myth acceptance was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Rape Myth Acceptance | Change from baseline in rape myth acceptance to up to eight months
  A revised version of the Illinois Rape Myth Acceptance Scale (Payne, Lonsway, & Fitzgerald, 1999) was used. The revised version (McMahon & Farmer, 2011) was selected because the scale includes updated language for college students as well as having a specific focus on accountability for rape and victim blaming (for information on scale development, see McMahon & Farmer, 2011). Students' rape myth acceptance was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011.
Rape Myth Acceptance | Change from baseline in rape myth acceptance to up to fifteen months
  A revised version of the Illinois Rape Myth Acceptance Scale (Payne, Lonsway, & Fitzgerald, 1999) was used. The revised version (McMahon & Farmer, 2011) was selected because the scale includes updated language for college students as well as having a specific focus on accountability for rape and victim blaming (for information on scale development, see McMahon & Farmer, 2011).Students' rape myth acceptance was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Rape Myth Acceptance | Change from baseline in rape myth acceptance to up to twenty months
  A revised version of the Illinois Rape Myth Acceptance Scale (Payne, Lonsway, & Fitzgerald, 1999) was used. The revised version (McMahon & Farmer, 2011) was selected because the scale includes updated language for college students as well as having a specific focus on accountability for rape and victim blaming (for information on scale development, see McMahon & Farmer, 2011).Students' rape myth acceptance assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.
Proclivity to Perpetrate Sexual Violence | Change from baseline in proclivity to perpetrate sexual violence to up to three months
  For proclivity to perpetrate, we used an item from Malamuth's (1989) Attraction to Sexual Aggression Scale and we created a question that combined items from Malamuth's scale and Lisak's Perpetrator History (PH) Scale (2000). These measures were assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Proclivity to Perpetrate Sexual Violence | Change from baseline in proclivity to perpetrate sexual violence to up to six months
  For proclivity to perpetrate, we used an item from Malamuth's (1989) Attraction to Sexual Aggression Scale and we created a question that combined items from Malamuth's scale and Lisak's Perpetrator History (PH) Scale (2000). These measures were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Proclivity to Perpetrate Sexual Violence | Change from baseline in proclivity to perpetrate sexual violence to up to eight months
  For proclivity to perpetrate, we used an item from Malamuth's (1989) Attraction to Sexual Aggression Scale and we created a question that combined items from Malamuth's scale and Lisak's Perpetrator History (PH) Scale (2000). These measures were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Proclivity to Perpetrate Sexual Violence | Change from baseline in proclivity to perpetrate sexual violence up to fifteen months
  For proclivity to perpetrate, we used an item from Malamuth's (1989) Attraction to Sexual Aggression Scale and we created a question that combined items from Malamuth's scale and Lisak's Perpetrator History (PH) Scale (2000). These measures were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Proclivity to Perpetrate Sexual Violence | Change from baseline in proclivity to perpetrate sexual violence to up to twenty months
  For proclivity to perpetrate, we used an item from Malamuth's (1989) Attraction to Sexual Aggression Scale and we created a question that combined items from Malamuth's scale and Lisak's Perpetrator History (PH) Scale (2000). These measures were assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.
Sexual Violence Perpetration | Change from baseline in sexual violence perpetration to up to three months
  Two questions from Lisak's Perpetrator History (PH) Scale (Lisak, Conklin, Hopper, Miller, Altschuler & Smith, 2000) were used to assess actual perpetration. Students' past perpetration was assessed via (1) a paper survey in June, July or August 2010 (baseline) and (2) a follow-up web-based survey in early September, 2010. All study participants received one dose of the intervention in June, July or August.
Sexual Violence Perpetration | Change from baseline in sexual violence perpetration to up to six months
  Two questions from Lisak's Perpetrator History (PH) Scale (Lisak, Conklin, Hopper, Miller, Altschuler & Smith, 2000) were used to assess actual perpetration. Students' past perpetration was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; and (3) a follow-up web-based survey in early December 2010. After the September, 2010 follow-up survey, participants were randomized to either receive two additional doses in October, 2010 and November, 2010 (experimental group) or no additional doses (control group).
Sexual Violence Perpetration | Change from baseline in sexual violence perpetration to up to eight months
  Two questions from Lisak's Perpetrator History (PH) Scale (Lisak, Conklin, Hopper, Miller, Altschuler & Smith, 2000) were used to assess actual perpetration. Students' past perpetration was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; and (4) a follow-up web-based survey in February, 2011.
Sexual Violence Perpetration | Change from baseline in sexual violence perpetration to up to fifteen months
  Two questions from Lisak's Perpetrator History (PH) Scale (Lisak, Conklin, Hopper, Miller, Altschuler & Smith, 2000) were used to assess actual perpetration. Students' past perpetration was assessed via(1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; and (5) a follow-up web-based survey in September, 2011. After the September, 2011 survey, experimental group participants were randomized to receive one additional dose (a booster session) or no additional doses.
Sexual Violence Perpetration | Change from baseline in sexual violence perpetration to up to twenty months
  Two questions from Lisak's Perpetrator History (PH) Scale (Lisak, Conklin, Hopper, Miller, Altschuler & Smith, 2000) were used to assess actual perpetration. Students' past perpetration was assessed via (1) a paper survey in June, July or August 2010 (baseline); (2) a follow-up web-based survey in early September, 2010; (3) a follow-up web-based survey in early December 2010; (4) a follow-up web-based survey in February, 2011; (5) a follow-up web-based survey in September, 2011 and (6) a final follow-up web-based survey in February 2012.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah McMahon, PhD, Principal Investigator — Rutgers University School of Social Work; Judy Postmus, PhD, Principal Investigator — Rutgers University School of Social Work
Locations (1):
- Rutgers, the State University of New Jersey, New Brunswick, New Jersey, United States

REFERENCES:
- [Background] McMahon S, Allen CT, Postmus JL, McMahon SM, Peterson NA, Lowe Hoffman M. Measuring bystander attitudes and behavior to prevent sexual violence. J Am Coll Health. 2014;62(1):58-66. doi: 10.1080/07448481.2013.849258. PMID 24313697
- [Result] McMahon, S., Hoffman, M., McMahon, S.M., Zucker, S. & Koenick, R.A. (2013). What Would You Do? Strategies for Bystander Intervention to Prevent Sexual Violence by College Students. Journal of College and Character, 14(2), p.141-152.